CLINICAL TRIAL: NCT06743347
Title: Dynamic Measurement of Cerebrospinal Fluid in Healthy Subjects: Pilot Study
Acronym: DYNA-LCS P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-A02411-46
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Cerebrospinal Fluid; Healthy Subjects or Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Contrast MRI (Experimental)
  Interventions: Other: MRI Contrast

INTERVENTIONS:
Other: MRI Contrast — Pass a Phase Contrast MRI. No injection required.

SUMMARY:
This research will enhance our knowledge and understanding of Cerebrospinal Fluid (CSF) circulation around the Central Nervous System (CNS) (brain and spinal cord).

The main objective is to obtain flow velocities using Phase Contrast (PC) MRI over the entire subarachnoid space (SAS). This will enable us to develop and validate a numerical model of the SAS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of agreement
* Free subject, without guardianship or curatorship or subordination
* Patients benefiting from a Social Security scheme or benefiting from it through a third party
* Informed consent signed by the patient after clear and complete information about the study

Exclusion Criteria:

* 3T MRI contraindications (pacemaker, cochlear implant, metallic splinter, etc)
* History of neurological pathology
* Previous operations involving the central nervous system (spinal surgery, neurological surgery, etc.)
* Current pathology or treatment that may interfere with the CSF or subarachnoid spaces (CSF dysregulation, disc herniation, hydrocephalus, Chiari malformation, etc.)
* Concurrent participation in another clinical research study
* Persons not covered by Social Security or not covered by Social Security through a third party
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection
* Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception (hormonal/mechanical: oral, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy)

Exclusion criteria during the study:

- Discovery of a contraindication to 3T MRI (pacemaker, cochlear implant, metallic splinter, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-09-24 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the velocity displacement of CSF about 7 planes (intracranial plane, C2-C3, C5-C6, T4-T5, T10-T11, L3-L4, L5-S1) | Time PC-MRI will be around 60min
  Displacement velocities of CSF will be obtain by Phase Contrats MRI.

SECONDARY OUTCOMES:
Using morphological MRI to model a digital twin | Time PC-MRI will be around 60min
  Comparison of velocity fields for each measurement section plane
To evaluate the velocity displacement of blood about 2 planes (intracranial plane, C2-C3) | Time PC-MRI will be around 60min
  Displacement velocities of blood will be obtain by Phase Contrats MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided